CLINICAL TRIAL: NCT00968214
Title: A Genome-Wide Association Study in Patients Experiencing Musculoskeletal Adverse Events on NCIC CTG Trial MA.27 Evaluating Aromatase Inhibitors as Adjuvant Therapy in Early Breast Cancer. A Collaboration Between the NIH Pharmacogenetics Research Network and the RIKEN Yokohama Institute Center for Genomic Medicine.
Brief Title: Study of Tumor and Blood Samples From Postmenopausal Women With Primary Breast Cancer Enrolled on Clinical Trial CAN-NCIC-MA27
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-TBCI-MA.27A; NCCTG-TBCI-MA.27A; CDR0000600225 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00694 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: DNA from blood specimens that have been previously collected from patients are analyzed for single nucleotide polymorphisms.
  Interventions: Genetic: polymorphism analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tumor and blood samples from postmenopausal women with primary breast cancer enrolled on clinical trial CAN-NCIC-MA27.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify genetic variation, as measured by single nucleotide polymorphisms, that is associated with musculoskeletal adverse events in specimens from postmenopausal women with hormone receptor-positive primary breast cancer receiving adjuvant aromatase inhibitors and enrolled on clinical trial CAN-NCIC-MA27.

OUTLINE: This is a multicenter study.

DNA from tumor tissue and blood specimens that have been previously collected from patients are analyzed for single nucleotide polymorphisms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer

  * Complete resection of primary tumor
  * Stage I-III (T1-3, N0-3, M0) disease
* Enrolled in clinical trial CAN-NCIC-MA27.
* No locally recurrent or metastatic breast cancer
* Hormone receptor status:

  * Estrogen receptor- or progesterone receptor-positive disease

PATIENT CHARACTERISTICS:

* Postmenopausal status, defined as one of the following:

  * At least 60 years old
  * Age 45-59 years with spontaneous cessation of menses for > 12 months prior to chemotherapy or study randomization
  * Age 45-59 years with cessation of menses for < 12 months or secondary to hysterectomy AND a follicle-stimulating hormone (FSH) level in the postmenopausal range (or > 34.4 IU/L)
  * Age 45-59 years on hormone replacement therapy (HRT) and discontinued HRT at diagnosis of breast cancer AND FSH level in the postmenopausal range (or > 34.4 IU/L)
  * Bilateral oophorectomy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the MA.27 clinical trial who received either anastrozole or exemestane for adjuvant therapy of resected early breast cancer
Sampling Method: Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2008-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Genetic variation associated with musculoskeletal adverse events | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Ingle, MD, Study Chair — Mayo Clinic